CLINICAL TRIAL: NCT07012720
Title: Research on the Potential Mechanisms Underlying the Efficacy Differences in Specific Neoadjuvant Treatment Regimens for Different Subtypes of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KY20242085-C-1
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Single-cell sequencing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- TNBC-Chemotherapy combined with immunotherapy (Experimental): Patients with TNBC subtype breast cancer receive chemotherapy combined with immunotherapy
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- TNBC-Chemotherapy (Experimental): Patients with TNBC subtype breast cancer receive chemotherapy
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- TNBC-Immunotherapy (Experimental): Patients with TNBC subtype breast cancer receive immunotherapy
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- HER2+HR- -EC-THP chemotherapy combined with targeted therapy regimen (Experimental): Patients with HER2+HR- subtype breast cancer receive EC-THP chemotherapy combined with targeted therapy
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- HER2+HR -- HP targeted treatment regimen (Experimental): Patients with HER2+HR- subtype breast cancer receive HP-targeted therapy regimens
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- HER2-HR+-AI+CDK4/6i Endocrine combined with CDK4/6 inhibitor regimen (Experimental): Patients with HER2-HR+ breast cancer were given a treatment regimen of endocrine combined with CDK4/6 inhibitors
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome
- HER2-HR+-AI Endocrine inhibitor regimen (Experimental): Endocrine therapy regimens were given to patients with HER2-HR+ breast cancer
  Interventions: Diagnostic Test: Single-cell sequencing and spatial transcriptome

INTERVENTIONS:
Diagnostic Test: Single-cell sequencing and spatial transcriptome — Tumor tissue samples of all enrolled patients before and after neoadjuvant therapy were collected. Based on single-cell sequencing and spatial transcriptome technology, the transcriptomic differences in neoadjuvant therapy response or treatment resistance under the same treatment regimen, as well as the transcriptomic changes of tumor tissues before and after treatment were explored.

SUMMARY:
This study is a single-center, open-label, prospective, clinical cohort study. It enrolled patients in three subgroups: triple negative, HR+HER2-, or HR-HER2+ subtypes, who will receive neoadjuvant treatment according to guidelines. Patients in each subgroup will be divided into two categories: those responsive to neoadjuvant therapy and those resistant to it, based on the efficacy of the treatment. Tumor tissue samples from all enrolled patients before and after neoadjuvant therapy will be collected. We will explore transcriptomic differences in neoadjuvant therapy responders or resisters under the same treatment regimen, as well as transcriptomic changes in tumor tissue before and after treatment, based on single-cell sequencing and spatial transcriptomic technology.

DETAILED DESCRIPTION:
This single-center, open, prospective, clinical cohort study plan recruited 71 patients with three subtypes of breast cancer: triple-negative type, HR+HER2-, and HR-HER2+. Based on the basic conditions of the enrolled patients, such as tumor stage, pathological classification, expression levels of tumor biomarkers, age and economic status of the patients, treatment plans suitable for the patients were formulated by referring to the recommended treatment methods for each subtype of breast cancer clearly stated in the 2023 edition of the CSCO Breast Cancer Diagnosis and Treatment Guidelines. Patients with triple-negative breast cancer: Group A received neoadjuvant chemotherapy combined with anti-PD1 immunotherapy (T-EC regimen combined with anti-PD1 treatment), Group B received neoadjuvant chemotherapy (T-EC regimen), and Group C received neoadjuvant anti-PD1 immunotherapy (patients explicitly refused chemotherapy). Based on the evaluation results of imaging efficacy before and after neoadjuvant therapy, patients in groups A and B were divided into two subgroups: treatment response and treatment resistance. Among them, 6 cases were selected from each of the two subgroups in group A for single-cell sequencing analysis. In Group B, 3 cases were selected from each of the two subgroups for single-cell sequencing analysis; Group C was expected to have a smaller population and no distinction was made regarding the therapeutic effect. Three cases were selected for single-cell sequencing analysis. Patients with HER2+HR- breast cancer: Group A received neoadjuvant chemotherapy combined with trastuzumab plus pertuzumab targeted therapy (EC-THP regimen), and Group B received neoadjuvant trastuzumab plus pertuzumab targeted therapy (HP regimen) (patients explicitly refused chemotherapy). Based on the preoperative imaging efficacy evaluation results of the patients in each treatment group, the patients were divided into two subgroups: treatment response and treatment resistance. Among them, 3 cases were selected from each of the two subgroups in group A for single-cell sequencing analysis, and 3 cases were selected from each of the two subgroups in Group B for single-cell sequencing analysis. Patients with HER2-HR+ breast cancer: Group A received neoadjuvant aromatase inhibitor combined with CDK4/6 inhibitor treatment (AI+CDK4/6i regimen), and Group B received neoadjuvant aromatase inhibitor treatment (AI monotherapy regimen). Based on the preoperative imaging efficacy evaluation results of the patients in each treatment group, the patients were divided into two subgroups: treatment response and treatment resistance. Three cases were selected from each subgroup of Group A and Group B for single-cell sequencing analysis.

Inclusion criteria:

1) Voluntary enrollment, able to understand and sign the informed consent form; 2) Female, aged 25 to 70; 3) Meet the indications for neoadjuvant therapy (based on the indicated population clearly defined in the 2023 CSCO Breast Cancer Diagnosis and Treatment Guidelines); 4) No previous systemic treatment for breast cancer; 5) The neoadjuvant treatment regimen met the inclusion requirements: triple-negative breast cancer (T-EC+antiPD-1/T-EC/antiPD-1) HER2+ HR-breast cancer (EC-THP/HP), HER2-HR+ breast cancer (AI/AI+CDK4/6i); 6) Tumor specimens can be obtained (including puncture, minimally invasive, incision biopsy, and surgery); 7) A complete pathological report can be obtained. 4.2 Exclusion Criteria:

1. The patient did not sign the informed consent form;
2. Tumor specimens cannot be obtained (including puncture, minimally invasive, incision biopsy, and surgery);
3. Patients with severe systemic infections or accompanied by other serious diseases;
4. Have received cytotoxic chemotherapy, endocrine therapy, biological therapy or radiotherapy for any previous reason;
5. Does not meet the indications for neoadjuvant therapy;
6. Neoadjuvant treatment regimens are not included in the neoadjuvant treatment regimens defined in this study;
7. Other circumstances where the researcher deems it unsuitable for inclusion. 4.3 Criteria for Subjects to withdraw from the study (1) All subjects can voluntarily withdraw at any stage of the study without being discriminated against or retaliated against, and their medical treatment will not be affected.

(2) Furthermore, the subjects may withdraw from this study under the following circumstances:

1. Withdrawal decided by the researcher:

   A: The patient does not meet the indications for the above-mentioned designated neoadjuvant regimen; B: In cases where the subjects are not suitable to continue the trial during the research process, such as when the patients cannot tolerate immunotherapy or chemotherapy, the established neoadjuvant treatment plan needs to be terminated; C: Those who accept the neoadjuvant treatment regimen specified in this study and show disease progression in the cycle evaluation need to terminate the neoadjuvant treatment in advance and undergo surgical resection of the tumor tissue.

   D: Adverse events occurred. It was judged by the researchers that continuing to participate in the study would have an adverse impact on the safety of the subjects.

   E: Subjects with poor compliance, which affects the assessment of tolerance; F: The researcher requests the subjects to withdraw from the study for any medical reason; G: The researchers believe that the subjects have other circumstances that make them unsuitable to continue participating in the trial.
2. Voluntary withdrawal of the subjects:

A: The subject was unwilling to continue participating in the study and voluntarily withdrew the informed consent form.

B: Loss to follow-up (Before loss to follow-up, subjects who have completed three visits should be attempted to be contacted).

ELIGIBILITY:
Inclusion criteria:

1. Voluntary enrollment, able to understand and sign the informed consent form;
2. Female, aged 25 to 70;
3. Meet the indications for neoadjuvant therapy (based on the indicated population clearly defined in the 2023 CSCO Breast Cancer Diagnosis and Treatment Guidelines);
4. No previous systemic treatment for breast cancer;
5. The neoadjuvant treatment regimen met the inclusion requirements: triple-negative breast cancer (T-EC+antiPD-1/T-EC/antiPD-1) HER2+ HR-breast cancer (EC-THP/HP), HER2-HR+ breast cancer (AI/AI+CDK4/6i);
6. Tumor specimens can be obtained (including puncture, minimally invasive, incision biopsy, and surgery);
7. A complete pathological report can be obtained.

Exclusion Criteria:

1. The patient did not sign the informed consent form;
2. Tumor specimens cannot be obtained (including puncture, minimally invasive, incision biopsy, and surgery);
3. Patients with severe systemic infections or accompanied by other serious diseases;
4. Have received cytotoxic chemotherapy, endocrine therapy, biological therapy or radiotherapy for any previous reason;
5. Does not meet the indications for neoadjuvant therapy;
6. Neoadjuvant treatment regimens are not included in the neoadjuvant treatment regimens defined in this study;
7. Other circumstances where the researcher deems it unsuitable for inclusion. Criteria for Subjects to withdraw from the study (1) All subjects can voluntarily withdraw at any stage of the study without being discriminated against or retaliated against, and their medical treatment will not be affected.

(2) Furthermore, the subjects may withdraw from this study under the following circumstances:

1. Withdrawal decided by the researcher:

   A: The patient does not meet the indications for the above-mentioned designated neoadjuvant regimen; B: In cases where the subjects are not suitable to continue the trial during the research process, such as when the patients cannot tolerate immunotherapy or chemotherapy, the established neoadjuvant treatment plan needs to be terminated; C: Those who accept the neoadjuvant treatment regimen specified in this study and show disease progression in the cycle evaluation need to terminate the neoadjuvant treatment in advance and undergo surgical resection of the tumor tissue.

   D: Adverse events occurred. It was judged by the researchers that continuing to participate in the study would have an adverse impact on the safety of the subjects.

   E: Subjects with poor compliance, which affects the assessment of tolerance; F: The researcher requests the subjects to withdraw from the study for any medical reason; G: The researchers believe that the subjects have other circumstances that make them unsuitable to continue participating in the trial.
2. Voluntary withdrawal of the subjects:

A: The subject was unwilling to continue participating in the study and voluntarily withdrew the informed consent form.

B: Loss to follow-up (Before loss to follow-up, subjects who have completed three visits should be attempted to be contacted).

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
RECIST1.1 Evaluates clinical efficacy | At 24 weeks
  At the end of neoadjuvant therapy, based on the preoperative MRI imaging results, the clinical efficacy was evaluated according to the Response Evaluation Criteria (RECIST1.1) for Solid tumors: complete response (CR) or partial response (PR), stable disease (SD) or disease progression (PD). The efficacy of neoadjuvant therapy was set as the primary endpoint of the study.

SECONDARY OUTCOMES:
residual cancer burden（RCB） | Two weeks after the operation
  The RCB score proposed by MD Anderson Cancer Center is a scoring standard based on the pathological specimens of the tumor bed and regional lymph nodes after breast cancer surgery and the results of microscopic sections. The RCB score and classification can be obtained using a calculator. This score comprehensively analyzed the two-dimensional size of the maximum residual tumor bed, the proportion of tumor cells and in situ cancer cells, as well as the number of positive lymph nodes and tumor metastasis. By adjusting the above variables and combining them with weighting factors, a continuous scoring method was formed to predict the prognosis of breast cancer patients with NACT. Among them, the maximum residual tumor bed is defined as the area where tumor cells are distributed under the microscope, while the cytological characteristics of breast cancer are obtained by evaluating the proportion of tumor cells and in situ cancer cells in the maximum tumor bed through microscopic sections
Pathological complete response (pCR) | Two weeks after the operation
  Pathological complete response generally refers to the situation where no histological evidence of malignant tumor can be found in the primary lesion of the breast, or only the component of carcinoma in situ remains. Strictly speaking, it refers to the fact that both the primary lesion of the breast and the metastatic regional lymph nodes have achieved pCR.
Disease-free survival (DFS) | Greater than or equal to 5 years after the operation.
  Disease-free survival (DFS) refers to the time from the start of randomization to disease recurrence or the death of patients due to disease progression. This trial requires that the postoperative follow-up period be greater than or equal to 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided